# **COVER PAGE**

# **Study Protocol**

The Effect of Ophiocephalus striatus Extract on IGF-1 and IL-6

Levels in Elderly Patients with Sarcopenia

**Trial Registration Number:** NCT05869383

**Date of document:** 15 March 2023

**Study Objective:** To investigate the effects of Ophiocephalus striatus extract on insulin-like growth factor-1 serum, interleukin-6 serum levels, and sarcopenia-related parameters in older adults with sarcopenia.

#### **Study Design:**

- Double-blind, randomized controlled trial.
- 80 older adults with sarcopenia.
- Intervention: Ophiocephalus striatus extract or placebo for two weeks.
- Primary outcomes: IGF-1 serum and IL-6 serum levels.

## **Study Methods:**

#### • Participants:

- o Inclusion criteria: Older adults (≥60 years old) with sarcopenia diagnosed using AWGS criteria.
- Exclusion criteria: Patients with severe chronic liver disease, impaired kidney function, acute disease phase, malignancy, depression, history of hypersensitivity to Ophiocephalus striatus, or those who refused to participate.

#### • Intervention:

- o Ophiocephalus striatus extract (5 g twice daily) or placebo for 2 weeks.
- o Both groups received a tailored diet.

#### • Data Collection:

Sociodemographic information, comorbidities, physical examinations, anthropometric measurements, nutrition assessment, functional status assessment, mental status assessment, cognitive status assessment, sarcopenia screening, handgrip strength assessment, 6 m walk speed assessment, muscle mass assessment, laboratory tests for IGF-1 and IL-6.

#### • Outcome Measures:

- o Primary outcomes: IGF-1 and IL-6 serum levels.
- Secondary outcomes: Calf circumference, appendicular skeletal muscle mass index (ASMI), handgrip strength, gait speed, creatinine levels.

#### • Data Processing and Analysis:

- o Descriptive and inferential statistics.
- o Paired t-tests, independent t-tests, Wilcoxon test, Mann-Whitney U tests.
- o p-value < 0.05 considered statistically significant.

#### **Study Results:**

- Significant reduction in serum IL-6 levels in the intervention group.
- Non-significant increase in IGF-1 levels in the intervention group.

• Improvements observed in calf circumference, ASMI, handgrip strength, and gait speed in the intervention group.

### **Study Conclusions:**

- Ophiocephalus striatus extract positively impacts serum IL-6 levels in older adults with sarcopenia.
- The study suggests that Ophiocephalus striatus extract may offer a valuable intervention for managing sarcopenia.

#### **Additional Notes:**

- The study was conducted at the Geriatric Clinic of RSUP Dr. Mohammad Hoesin, Palembang.
- Ethical clearance was obtained from the Research Ethics Commission (No. DP.04.03/D.XVIII.6.11/ETIK/36/2023).
- The study was conducted from March 2023 to August 2023.